CLINICAL TRIAL: NCT04589078
Title: Polyp REcognition Assisted by a Device Interactive Characterization Tool - The PREDICT Study
Acronym: PREDICT
Status: Completed | Type: Observational
Sponsor: Cosmo Artificial Intelligence-AI Ltd (Industry)
Responsible Party: Sponsor
Organization: Cosmo Pharmaceuticals NV (Industry)
Other Study IDs: CB-17-08/05
Record Dates: First submitted 2020-10-13; First posted 2020-10-19 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Artificial Intelligence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Interficial Intelligence: Each patient will undergo standard white-light colonoscopy with the support of the latest version of the CE marked GI Genius CADe available.
  Interventions: Device: GI Genius CADe system

INTERVENTIONS:
Device: GI Genius CADe system — Each patient will undergo standard white-light colonoscopy with the support of the latest version of the CE marked GI Genius CADe available.

SUMMARY:
Diminutive colorectal polyps (≤ 5 mm) represent most of the polyps detected during colonoscopy, especially in the rectum-sigmoid tract. The characterization of these polyps by virtual chromoendoscopy is recognized as a key element for innovative imaging techniques. As a matter of facts diminutive colorectal polyps are very frequent and, if located in the rectosigmoid colon, they present a very low malignant risk (0.3% of evolution towards advanced adenoma and up to 0.08% of evolution towards invasive carcinoma). The real-time characterization would allow to identify the lowest risk polyps (hyperplastic subtype), to leave them in situ or, if resected, not to send them for histological examination, allowing a huge saving in healthcare associated costs.

Recently, the American Society for Gastrointestinal Endoscopy (ASGE) Technology Committee established the Preservation and Incorporation of Valuable endoscopic Innovations (PIVI) document, specific for real-time histological assessment for tiny colorectal polyps, to establish reference quality thresholds. Two performance standards have been developed to guide the use of advanced imaging:

1. for diminutive polyps to be resected and discarded without pathologic assessment, endoscopic technology (when used with high confidence) used to determine histology of polyps ≤ 5mm in size, when combined with the histopathology assessment of polyps > 5 mm in size, should provide a ≥ 90% agreement in assignment of post-polypectomy surveillance intervals when compared to decisions based on pathology assessment of all identified polyps;
2. in order for a technology to be used to guide the decision to leave suspected rectosigmoid hyperplastic polyps ≤ 5 mm in size in place (without resection), the technology should provide ≥ 90% negative predictive value (when used with high confidence) for adenomatous histology.

Computer-Aided-Diagnosis (CAD) is an artificial intelligence-based tool that would allow rapid and objective characterization of these lesions. The GI Genius CADx was developed to help endoscopists in their clinical practices for polyps characterization.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 40-80 undergoing screening colonoscopy for CRC
* Ability to provide written, informed consent (approved by EC) and understand the responsibilities of trial participation.

Exclusion Criteria:

* subjects positive to Fecal Immunochemical Test or Fecal Occult Blood Test;
* subjects undergoing CRC surveillance colonoscopy
* subject at high risk for CRC
* subjects with a personal history of CRC, IBD or hereditary polyposic or non-polyposic syndromes;
* patients with previous resection of the sigmoid rectum;
* patients on anticoagulant therapy, which precludes resection / removal operations due to histopathological findings;
* patients who perform an emergency colonoscopy.

Ages: 40 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients aged 40-80 undergoing colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2020-12-22 (Actual)

PRIMARY OUTCOMES:
Negative Predictive Value of histology prediction on diminutive (≤5 mm) rectosigmoid polyps | 1 day

SECONDARY OUTCOMES:
Agreement in assignment of post-polypectomy surveillance intervals | 1 day
  Agreement in assignment of post-polypectomy surveillance intervals according to established guidelines between:
  * the assignment identified according to the combined
    * GI Genius CADx histology prediction for diminutive (≤5 mm) polyps and
    * histology for larger polyps (> 5 mm), and
  * the assignment identified according to histology only.

OTHER OUTCOMES:
Sensitivity, Specificity, Accuracy, PPV and NPV of GI Genius CADx histology prediction and endoscopist assessment on all the identified lesions | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Endoscopy Unit, Humanitas Research Hospital, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: No